CLINICAL TRIAL: NCT06434948
Title: The Effect of Omega 3 Supplementation on Postoperative Delirium in Elderly Patients Undergoing Major Cardiac Surgery: a Prospective, Randomized, Controlled Trial
Brief Title: The Effect of Omega 3 Supplementation on Postoperative Delirium in Elderly Patients Undergoing Major Cardiac Surgery
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Quinn Johnson, Department Chair of Anesthesiology and Perioperative Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2099184
Record Dates: First submitted 2024-05-09; First posted 2024-05-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; delirium; fish oil; omega 3; Lovaza; cardiac bypass; omega 3 ethyl esters
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Omacor

STUDY DESIGN:
Intervention Model Description: Arm 1: 4 grams of Omega-3 Ethyl Esters Arm 2: 2 grams of Omega-3 Ethyl Esters Arm 3: Standard of care
Masking Description: This study will not be blinded as there is no suitable placebo for omega-3 ethyl esters available at this time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Omega-3 Ethyl Esters 4 g (Experimental): Patients will be given 4 grams of omega-3 ethyl esters orally before surgery and for 3 days postoperatively.
  Interventions: Drug: Omega-3 Ethyl Esters 4 g
- Omega-3 Ethyl Esters 2 g (Experimental): Patients will be given 2 grams of omega-3 ethyl esters orally before surgery and for 3 days postoperatively.
  Interventions: Drug: Omega-3 Ethyl Esters 2 g
- Standard of Care (No Intervention): Patients will not receive any study drug.

INTERVENTIONS:
Drug: Omega-3 Ethyl Esters 4 g — 4 grams = 4 capsules, once daily
  Other Names: Omega-3 ethyl esters; Lovaza
  Arms: Omega-3 Ethyl Esters 4 g
Drug: Omega-3 Ethyl Esters 2 g — 2 grams = 2 capsules, once daily
  Other Names: Lovaza; Omega-3 ethyl esters
  Arms: Omega-3 Ethyl Esters 2 g

SUMMARY:
The purpose of this study is to determine whether giving omega-3 fatty acids prior to and after cardiac bypass surgeries decreases the incidence of postoperative delirium in patients aged 65 and over.

DETAILED DESCRIPTION:
Patients aged 65 years and over requiring elective cardiac bypass surgeries will receive either 0, 2, or 4 grams of omega-3 ethyl esters before their surgery and for 3 days postoperatively to determine whether there is an affect on the incidence of postoperative delirium. All patients will receive hospital standard of care therapy for their surgery and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* American Society of Anesthesiologists (ASA) Class Physical Status I-IV

Exclusion Criteria:

* Inability to obtain written informed consent.
* Inability to take study drug due to intubation or other reason.
* Delirium present at screening.
* Known hypersensitivity (e.g. anaphylactic reaction) to omega-3 ethyl esters or any of its components
* Allergy to fish or shellfish
* Currently taking warfarin (Coumadin), apixaban (Eliquis), dabigatran (Pradaxa), edoxaban (Savaysa/Lixiana), rivaroxaban (Xarelto), or other anticoagulant drugs.
* Currently taking omega-3, omega-6, vitamin E, or fish oil supplements.
* Significant renal disease with a serum creatinine ≥ 2 mg/dL.
* Significant liver disease with alanine aminotransferase (ALT) levels 1.5 times the normal range of 6-45 units/liter and aspartate transferase (AST) levels 1.5 times the normal range of 10-42 units/liter.
* History or diagnosis of diabetes.
* History or diagnosis of neurodegenerative disease such as Parkinson's, Alzheimer's, or dementia.
* History or diagnosis of bleeding disorder.
* History or diagnosis of metabolic syndrome or disorder.
* History or diagnosis of thyroid problems such as hyperthyroidism or hypothyroidism.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Presence of Postoperative Delirium | From the date of surgery until the patient is discharged, up to 30 days.
  Number of patients that experienced postoperative delirium during the study.

SECONDARY OUTCOMES:
Postoperative Delirium Symptoms | From the date of surgery until the patient is discharged, up to 30 days.
  Presence of any postoperative delirium symptoms during patient's hospital stay.
Length of Stay | From the date of surgery until the patient is discharged, up to 30 days.
  Number of days patient stayed in hospital from the time of admission to discharge.
Type of Anesthesia Used | During surgery, up to 24 hours
  Number of patients administered anesthesia using mainly propofol or sevoflurane.
Amount of Pain Medication Given Postoperatively | From the date of surgery until the patient is discharged, up to 30 days.
  Average morphine milligram equivalents given to patients postoperatively until their discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Quinn Johnson, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No